CLINICAL TRIAL: NCT04755400
Title: The Effect of Orally Administrated Nitrate on Renal Parameters and Systemic Haemodynamics, in a Randomized, Placebo Controlled, Crossed Over Study on Healthy Subjects.
Brief Title: The Effect of Orally Administrated Nitrate on Renal Parameters and Systemic Haemodynamics
Acronym: APNI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frank Mose (Other)
Collaborators: Herning Hospital (Other)
Responsible Party: Sponsor-Investigator, Frank Mose, Associate professor, Region MidtJylland Denmark
Organization: Region MidtJylland Denmark (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AMH-1-2016
Record Dates: First submitted 2021-02-03; First posted 2021-02-16 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — potassium nitrate; Potassium Chloride

STUDY DESIGN:
Intervention Model Description: double-blinded, placebo-controlled, crossover study
Who Masked: Participant, Care Provider, Investigator
Masking Description: The Hospital Pharmacy, Herning Hospital, generates the randomization list. A copy of the list is kept at the Medical Research department.
  Patients are randomized to receive either potassium nitrate or placebo (Potassium chloride). The Hospital Pharmacy, Gødstrup Hospital, will blind both treatments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potassium Nitrate (Active Comparator): 4 days treatment with 24 mmol potassium nitrate capsules
  Interventions: Other: isotonic saline 9%; Dietary Supplement: Potassium nitrate
- Potassium Chloride (Placebo Comparator): 4 days treatment 24 mmol potassium chloride capsules
  Interventions: Other: isotonic saline 9%; Dietary Supplement: Potassium chloride

INTERVENTIONS:
Other: isotonic saline 9% — 1 Liter of Isotonic saline administered I.V.
  Other Names: Sodium Chloride 9%
Dietary Supplement: Potassium nitrate — 24 mmol of Potassium nitrate is the active comparator substance, that is ingested every morning for 4 days before and on the examination day.
  Arms: Potassium Nitrate
Dietary Supplement: Potassium chloride — 24 mmol of Potassium nitrate is the placebo substance, that is ingested every morning for 4 days before and on the examination day.
  Arms: Potassium Chloride

SUMMARY:
Treatment with nitrate has shown to lower blood pressure in both healthy subjects and hypertensive patients.Beside this nitrate have also shown to decrease arterial stiffness and improve endothelial function.But the effect of nitrate on renal blood flow, kidney function, water and salt balance and vasoactive hormones is still unclear.

Therefore, the purpose of this study is to investigate the effect of orally administered nitrate on these parameters.

This will be done in a double-blinded, placebo-controlled, crossover study. 20 healthy subjects will be treated, in a randomized order, with both potassium nitrate and placebo separated by at least 4 weeks wash-out.

DETAILED DESCRIPTION:
Inorganic nitrate reduces blood pressure and improves endothelial function in both healthy subjects and hypertensive patients.

This effect is thought to be caused through bioconversion to nitric oxide. Thus improving risk factors of cardiovascular decease by increasing vasodilatation, salt regulation and vasoactive hormones.The purpose of this study is to investigate the effect of inorganic nitrate on kidney function, hormones and circulation, which is still unknown.

The effect of 4 days treatment with 24 mmol potassium nitrate capsules on heart rate, blood pressure, vasoactive hormones and urinary excretion of sodium and water will be measured in a randomized, placebo controlled, double blinded, crossover study in 20 healthy subjects. Each subject attends 2x2 examination days at least 4 weeks apart. The examination days are divided into 8 clearance periods of 30 min. each. The first 3 are baseline periods and in period 4 1 Liter of saline is administered to detect any difference in renal parameters after NaCl load.

If inorganic nitrate supplementation is found to lower blood pressure in addition to favorable renal effects, it could lead to changes in the general treatment of high blood pressure and cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64 years
* BMI 18,5-30
* Normotensive
* Women must use contraception

Exclusion Criteria:

* Tobacco smoking (Non-smokers in more than 3 months can be included)
* Medicine- or drug abuse
* Alcohol abuse >7 units for women >14 units for men
* Medical treatment (over the counter medication will evaluated whether or not it is grounds for exclusion) within 2 weeks before the trail period starts except contraception.
* Pregnancy or nursing
* Neoplastic disorders
* Significant clinical signs of heart-, lung-, liver-, kidney-, endocrine- or brain disorders
* Clinically significant abnormal findings in screening blood samples, urine sample or ECG - Donation of blood within 1 month of the first day of investigation.
* Allergy against compounds in investigational medicine

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Glomerular filtration rate (GFR) | analysed right after each examination day. (day 1)
  mL/minute

SECONDARY OUTCOMES:
Brachial blood pressure (BP) | analysed right after each examination day. (day 1)
  mmhg
central blood pressure (cSBP) | analysed right after each examination day. (day 1)
  mmhg
Heart rate | analysed right after each examination day. (day 1)
  beats pr. min.
Pulse wave velocity (PWV) | analysed right after each examination day. (day 1)
  measured via Mobilograph
Total vascular resistance (TVR) | analysed right after each examination day. (day 1)
  measured via Mobilograph
Augmentation index (Aix@75) | analysed right after each examination day. (day 1)
  measured via Mobilograph
Urinary excretions of aquaporin-2 (u-AQP2) | Centrifuged and hereafter frozen. Analyzed during the following 12 months.
  ng/mmol crea
Urinary excretions of epithelial sodium channels (u-ENaCγ) | Centrifuged and hereafter frozen. Analyzed during the following 12 months.
  ng/mmol crea
Urinary excretions of Na-Cl cotransporter (u-NCC). | Centrifuged and hereafter frozen. Analyzed during the following 12 months.
  ng/mmol crea
plasma concentration of renin (PRC) | Centrifuged and hereafter frozen. Analyzed during the following 12 months.
  pg/mL
plasma concentration of angiotensin II (p-AngII) | Centrifuged and hereafter frozen. Analyzed during the following 12 months.
  pg/mL
plasma concentration of aldosterone (p-Aldo) | Centrifuged and hereafter frozen. Analyzed during the following 12 months.
  pmol/L
plasma concentration of arginine vasopressin (p-AVP) | Centrifuged and hereafter frozen. Analyzed during the following 12 months.
  pg/mL
plasma concentration of atrial natriuretic peptide (p-ANP) | Centrifuged and hereafter frozen. Analyzed during the following 12 months.
  pmol/L
plasma concentration of brain natriuretic peptide (p-BNP). | Centrifuged and hereafter frozen. Analyzed during the following 12 months.
  pmol/L
plasma and urine levels of Nitrate (NO3) | Centrifuged and hereafter frozen. Analyzed during the following 12 months.
  μmol/L
plasma and urine levels of nitrite (NO2) | Centrifuged and hereafter frozen. Analyzed during the following 12 months.
  μmol/L
plasma and urine levels of cyclic guanosine monophosphate (cGMP). | Centrifuged and hereafter frozen. Analyzed during the following 12 months.
  pmol/mL
Creatinine clearance (CrCl) | analysed right after each examination day. (day 1)
  mL/minute
Urinary excretion rate of sodium (U-Na) | analysed right after each examination day. (day 1)
  mmol/min
Urinary excretion rate of potassium(U-K) | analysed right after each examination day. (day 1)
  mmol/min
Free water clearance (CH2O) | analysed right after each examination day. (day 1)
  mL/minute
Fractional excretion of sodium (FENa) | analysed right after each examination day. (day 1)
  calculated into %
Fractional excretion of potassium (FEK) | analysed right after each examination day. (day 1)
  calculated into %
Urinary excretion rate of albumin (UAER) | analysed right after each examination day. (day 1)
  µg/min

CONTACTS AND LOCATIONS:
Overall Officials: Jesper N Bech, Ph.D., M.D., Study Director — University of Aarhus
Locations (1):
- Godstrup Hospital, Herning, Denmark